CLINICAL TRIAL: NCT03699306
Title: Comparison of Three Methods for NG Tube Placement in Intubated Patients in the Emergency Department During 2016-2018
Brief Title: Comparison of Three Methods for NG Tube Placement
Acronym: NG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Principle investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 396780
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Unconsciousness
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional r blinded (Active Comparator): the participants were allocated to have NG tube inserted in a conventional or blind method.
  Interventions: Procedure: NG tube insertion method
- Brake cable (Active Comparator): the participants were assigned to have NG tube inserted by use of a bike brake cable as a guide wire.
  Interventions: Procedure: NG tube insertion method
- High way man's hitch (Active Comparator): they were selected to have NG tube inserted by use of silk thread knot.
  Interventions: Procedure: NG tube insertion method

INTERVENTIONS:
Procedure: NG tube insertion method — a feeding tube called naso-gastric or NG tube were inserted through nostril inside the stomach randomly by one of three methods mentioned earlier
  Other Names: NG tube placement technique

SUMMARY:
Background and Aim: Tubular feeding is used, in patients who cannot take food through their mouths, but the digestive system has the ability to digest food. This method is safe and affordable for the patient and results in maintaining the function of the digestive system and reducing the risk of infection and sepsis. The purpose of this study was to compare the three methods of the NG tube placement in intubated patients in the emergency department of university-affiliated hospitals of Isfahan from2016 to 2018.

Materials and Methods: This study was a randomized and prospective clinical trial. The statistical population of this study was all patients who had been referred to the emergency department of Al-Zahra and Ayatollah Kashani hospitals in Isfahan between2016and2018. The sample size was 25 in each group, and in total 75 subjects. The first group was NG tube insertion by the conventional method, the second group was using brake cable and the third group was embeddedby highwayman's hitch or draw hitch, using a silk thread. For all patients, demographic characteristics and possible complications were recorded. Finally, the data were analyzed using SPSS20 software at two statistical levels of descriptive and inferential.

ELIGIBILITY:
Inclusion Criteria:

* all intubated patients, referred to the emergency department

Exclusion Criteria:

* the presence of symptoms of skull base fracture,
* bleeding disorders and coagulopathies,
* maxillofacial trauma, which led to deformity and impairment of NG tube,
* upper respiratory tract diseases and anomalies,
* nasal congestion and nostril stenosis,
* esophageal disorder (esophageal stenosis and esophageal varicose vein),
* and a history of head and neck radiotherapy.
* Patients who had been intubated in other centers and being referred to these two centers were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
success rate | Intraoperative (time from entry of the NG tube through nostril til entering inside the stomach or whenever the operator declared.)
  success rate was defined as successfully inserted NG tube inside the stomach

SECONDARY OUTCOMES:
procedure duration | Intraoperative (from nostril entry til sromach entry or operatoe declaration as the end of procedure)
  it was measured as the total time from start of the procedure til the entry of the tube inside the stomach.

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Al-Zahra University Hospital, Isfahan
  - Mehdi Nasr Isfahani, Isfahan

IPD SHARING:
Plan to Share IPD: No